CLINICAL TRIAL: NCT03110029
Title: Evaluating the Efficacy and Compatibility of Efinaconazole 10% Solution (Jublia) for the Treatment of Toenail Onychomycosis in Patients Wearing Toenail Polish Compared to Those Without Polish
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Boni Elewski, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X141114004
Record Dates: First submitted 2015-10-16; First posted 2017-04-12 (Actual); Results first posted 2019-03-20 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Onychomycosis of Toenail
MeSH Terms: interventions — efinaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efinaconazole 10 % and Nail Polish (Active Comparator): Subject will have Efinaconazole 10% solution application and nail polish
  Interventions: Drug: Efinaconazole 10% Topical Application Solution [JUBLIA]; Other: Application of Nail Polish
- Efinaconazole 10% without Nail Polish (Placebo Comparator): Subject will have only Efinaconazole 10% application and no nail polish
  Interventions: Drug: Efinaconazole 10% Topical Application Solution [JUBLIA]

INTERVENTIONS:
Drug: Efinaconazole 10% Topical Application Solution [JUBLIA] — Topical efinaconazole 10% solution (Jublia)
  Other Names: Jublia
Other: Application of Nail Polish — Application of Nail Polish
  Arms: Efinaconazole 10 % and Nail Polish

SUMMARY:
This study will test how well efinaconazole solution (Jublia) works to treat toenail fungal infections in patients who wear polish compared to those who do not.

DETAILED DESCRIPTION:
Topical efinaconazole 10% solution is known to be an efficacious and safe treatment modality for toenail onychomycosis. This study will examine the compatibility of topical efinaconazole and nail polish in patients with distal and lateral subungual onychomycosis (DLSO). It is hypothesized that the treatment of DLSO with efinaconazole 10% solution will not be adversely affected by the application of nail polish.

ELIGIBILITY:
Inclusion Criteria:

* Female age 19-70, as 19 is the legal age in Alabama
* DLSO affecting at least 1 great toenail diagnosed with positive potassium hydroxide microscopy and culture of a dermatophyte
* Suitable for application of topical antifungal therapy, in the opinion of the investigator
* Target toenail thickness of 3 mm or less as measured by digital caliper, as thickness greater than 3 mm may allow inclusion of patient with severe onychomycosis, and this was the criteria used in the pivotal trial using topical efinaconazole for onychomycosis
* Women of childbearing potential will be required to use birth control and a negative urine pregnancy test must be documented prior to initiating treatment

Exclusion Criteria:

* History of immunosuppression or concurrent use of immunosuppressant drugs
* History of uncontrolled diabetes mellitus
* History of psoriasis or any other condition that might interfere with the toenail evaluation
* Three or more dermatophytomas (streaks) on the target nail
* Severe DLSO of the target nail
* Patients who cannot refrain from wearing gel or plastic based polishes that are used in salons and that require curing

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni E Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group (Frequently Wears Toenail Polish): Patients who self-identified as frequently wearing toenail polish were placed in the study group.
  Inclusion criteria consisted of being female and aged 19-70 with distal and lateral subungual onychomycosis (DLSO) effecting at least one great toenail. The target great toenail thickness was less than or equal to 3mm. DLSO was diagnosed by having a positive potassium hydroxide microscopy and culture of a dermatophyte. Exclusion criteria included a history of either immunosuppression, uncontrolled diabetes mellitus, or psoriasis. Patients were also excluded if they had severe target toenail DLSO or three or more dermatophytomas on the target toenail. Patients were required to refrain from wearing gel or plastic based polishes that are used in salons and require curing.
  Patients with symptomatic tinea pedis at screening were treated with luliconazole cream for 2 weeks.
- Control Group (no Toenail Polish): The control group was comprised of women who agreed to abstain from wearing toenail polish throughout the length of the study.
  Inclusion criteria consisted of being female and aged 19-70 with DLSO effecting at least one great toenail. The target great toenail thickness was less than or equal to 3mm. DLSO was diagnosed by having a positive potassium hydroxide microscopy and culture of a dermatophyte. Exclusion criteria included a history of either immunosuppression, uncontrolled diabetes mellitus, or psoriasis. Patients were also excluded if they had severe target toenail DLSO or three or more dermatophytomas on the target toenail. Patients were required to refrain from wearing gel or plastic based polishes that are used in salons and require curing.
  Patients with symptomatic tinea pedis at screening were treated with luliconazole cream for 2 weeks.
Period: Overall Study
Arm/Group | Study Group (Frequently Wears Toenail Polish) | Control Group (no Toenail Polish)
Started | 7 | 6
Completed | 6 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Wearing Toenail Polish: Subject will have Efinaconazole 10% application and nail polish
  Efinaconazole 10% (Jublia): Topical Efinaconazole 10% solution
  Application of nail polish
- Abstain From Wearing Toenail Polish: Subject will have Efinaconazole 10% application and no nail polish
  Efinaconazole 10% (Jublia): Topical Efinaconazole 10% solution
- Total: Total of all reporting groups
Arm/Group | Wearing Toenail Polish | Abstain From Wearing Toenail Polish | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Customized [Count of Participants; unit: Participants]
  19-70 | 7 | 6 | 13
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Not recorded | NA — Not recorded | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Nail Polish Disruption Using the Likert Scale
Description: Patients will answer the following question:
  Which will be answered using a Likert scale where 0 represents no alteration in polish and 10 represents complete destruction of the polish:
  Is the quality of your polish diminished with use of Jublia?
Time Frame: 52 weeks
Population: Only participants who completed the trial were included in results. Two participants withdrew due to personal scheduling conflicts.
Measure: Mean (Full Range); unit: percentage of nail polish disruption
Groups:
- Wearing Toenail Polish: Subject will have Efinaconazole 10% application and nail polish
  Efinaconazole 10% (Jublia): Topical efinaconazole 10% solution
  Application of nail polish: Application of nail polish only
Arm/Group | Wearing Toenail Polish | Abstain From Wearing Toenail Polish
Number analyzed (Participants) | 6 | 5
percentage of nail polish disruption | 0.6 [0 to 100] | 0 [0 to 100]

2. Secondary Outcome: Percentage of Disease Improvement Using Onychomycosis Severity Index (OSI)
Description: Using 3rd party blinding, DLSO was assessed at baseline and at every subsequent visit using the onychomycosis severity index (OSI), measuring percent of the target nail involved, and grading the infection from mild to moderate to severe. The range for OSI is 0-20 with 20 indicating severe nails disease. Nail growth was measured at each visit. Fungal testing was done at screening, 3 months, 7 months, end of treatment (48 weeks), and end of study (52 weeks). Clinical and mycologic cure was evaluated at week 52.
Time Frame: 52 week
Population: We did not include results from the two participants who withdrew from the study due to personal scheduling conflicts. Results for only 11 subjects who completed the study are represented in the number of participants analyzed.
Measure: Mean (Full Range); unit: percentage change target nail
Arm/Group | Wearing Toenail Polish | Abstain From Wearing Toenail Polish
Number analyzed (Participants) | 6 | 5
percentage change target nail | 0.56 [0 to 100] | 0.54 [0 to 100]

ADVERSE EVENTS:
Time Frame: 52 Weeks
Groups:
- Efinaconazole 10% and Nail Polish: Patients who self-identified as frequently wearing toenail polish were placed in the study group. Inclusion criteria consisted of being female and aged 19-70 with DLSO effecting at least one great toenail. The target great toenail thickness was less than or equal to 3mm. DLSO was diagnosed by having a positive potassium hydroxide microscopy and culture of a dermatophyte. Exclusion criteria included a history of either immunosuppression, uncontrolled diabetes mellitus, or psoriasis. Patients were also excluded if they had severe target toenail DLSO or three or more dermatophytomas on the target toenail. Patients were required to refrain from wearing gel or plastic based polishes that are used in salons and require curing.
  Patients with symptomatic tinea pedis at screening were treated with luliconazole cream for 2 weeks.
- Efinaconazole 10% Without Nail Polish: The control group was comprised of women who agreed to abstain from wearing toenail polish throughout the length of the study.
  Inclusion criteria consisted of being female and aged 19-70 with DLSO effecting at least one great toenail. The target great toenail thickness was less than or equal to 3mm. DLSO was diagnosed by having a positive potassium hydroxide microscopy and culture of a dermatophyte. Exclusion criteria included a history of either immunosuppression, uncontrolled diabetes mellitus, or psoriasis. Patients were also excluded if they had severe target toenail DLSO or three or more dermatophytomas on the target toenail. Patients were required to refrain from wearing gel or plastic based polishes that are used in salons and require curing.
  Patients with symptomatic tinea pedis at screening were treated with luliconazole cream for 2 weeks.
Arm/Group | Efinaconazole 10% and Nail Polish | Efinaconazole 10% Without Nail Polish
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03110029/Prot_SAP_000.pdf